CLINICAL TRIAL: NCT04244708
Title: Radiotherapy Plus Concomitant Temozolomide for Refractory Pituitary Adenomas，A Randomized，Double-blind, Placebo-controlled Phase II Trial
Brief Title: The Effect of Chemoradiotherapy in Patients With Refractory Pituitary Adenomas
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PekingUMCH-PA-TMZ
Record Dates: First submitted 2019-12-30; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pituitary Adenomas
Keywords: Temozolomide; radiotherapy; refractory pituitary adenomas
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy plus temozolomide (Experimental): Undergoing fractionated radiotherapy at a dose of 2 Gy per fraction given once daily five days per week for a total dose of 54 Gy, plus continuous daily temozolomide (75 mg per square meter of body-surface area per day), followed by six cycles of adjuvant temozolomide.
  Interventions: Drug: Radiotherapy plus temozolomide
- Radiotherapy plus placebo (Placebo Comparator): Radiotherapy treatment alone undergoing fractionated radiotherapy, total 54 Gy, 2GyX27, received placebo.
  Interventions: Other: Radiotherapy plus placebo

INTERVENTIONS:
Drug: Radiotherapy plus temozolomide — undergoing fractionated radiotherapy at a dose of 2 Gy per fraction given once daily five days per week (Monday through Friday) over a period of six weeks, for a total dose of 54 Gy, plus continuous daily temozolomide (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy), followed by six cycles of adjuvant temozolomide (150 to 200 mg per square meter for 5 days during each 28-day cycle).
  Arms: Radiotherapy plus temozolomide
Other: Radiotherapy plus placebo — undergoing fractionated radiotherapy at a dose of 2 Gy per fraction given once daily five days per week (Monday through Friday) over a period of six weeks, for a total dose of 54 Gy, plus placebo
  Arms: Radiotherapy plus placebo

SUMMARY:
The purpose of this study was to determine whether radiotherapy combined with Temozolomide is more effective than radiotherapy alone in the treatment of patients with refractory pituitary adenomas. The Basic treatment was Radiotherapy over a period of six weeks, for a total dose of 54 Gy. The150 participants were randomized to use either radiotherapy plus Temozolomide (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy), or radiotherapy plus placebo for 6 weeks. After a 4-week break, followed by six cycles of placebo or adjuvant temozolomide (150 to 200 mg per square meter for 5 days during each 28-day cycle). The primary end point was Objective Response rate, the second end point was PFS. Greater response was anticipated in patients treated with Temozolomide+ radiotherapy than radiotherapy alone.

DETAILED DESCRIPTION:
The purpose of this study was to determine whether radiotherapy combined with Temozolomide is more effective than radiotherapy alone in the treatment of patients with refractory pituitary adenomas. The Basic treatment was Radiotherapy, which is consisted of fractionated focal irradiation at a dose of 2 Gy per fraction given once daily five days per week (Monday through Friday) over a period of six weeks, for a total dose of 54 Gy. The150 participants were randomized to use either radiotherapy plus Temozolomide (75 mg per square meter of body-surface area per day, 7 days per week from the first to the last day of radiotherapy), or radiotherapy plus placebo for 6 weeks. After a 4-week break, patients were then to receive up to six cycles of adjuvant temozolomide or placebo according to the standard 5-day schedule every 28 days. The dose was 150 mg per square meter for the first cycle and was increased to 200 mg per square meter beginning with the second cycle, so long as there were no hematologic toxic effects followed by six cycles of placebo or adjuvant temozolomide (150 to 200 mg per square meter for 5 days during each 28-day cycle). The primary end point was Objective Response rate, the second end point was PFS. Greater response was anticipated in patients treated with Temozolomide+ radiotherapy than radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

Minimum Age: 18 Years Maximum Age: 80 Years

1. Age ≥18 years, regardless of gender;
2. Meet the diagnostic criteria for refractory pituitary tumors;

   1. The tumor showed invasive growth on imaging and rapid growth, Ki-67 labeling index ≥3%;
   2. The tumor recurred within a short period of time (< 6months) after total resection;
   3. The tumor continues to grow after surgery and medical therapy;
   4. Systemic examination showed no metastases in the cranial canal or other systems throughout the body.
3. Clinicopathological diagnosis of pituitary adenoma, and pathological tissue (wax or frozen tissue) can be obtained;
4. Expected survival time ≥ 6 months;
5. KPS score ≥70 points;
6. Subjects who were able to read, understand, and sign written informed consent prior to participating in the study and were willing to comply with protocol requirements.

Exclusion Criteria:

Participants cannot participate in this study if they meet any of the following conditions:

1. Subjects participated in clinical studies of other drugs or medical devices within 3 months before screening.
2. Known to be allergic to temozolomide capsules;
3. Have been diagnosed with pituitary carcinoma or have other malignant tumors;
4. Have received radiation therapy for Sella region;
5. Those with severe acute and chronic diseases in various systems, whose conditions have not been effectively controlled, and whose conditions are unstable, including but not limited to:

   1. Patients with cardiac insufficiency (NYHA cardiac function grade ≥ 2), patients with severe heart disease such as cardiomyopathy, coronary heart disease, severe arrhythmia, etc. that are not effectively controlled;
   2. Severe active infections,
   3. Uncontrollable diabetes, hypertension / hypotension, cerebrovascular disease, gastric ulcer, respiratory disease, active autoimmune disease, etc .;
   4. History of any other diseases that the researcher judges to be unsuitable for the trial, etc .;
6. For hepatic and renal insufficiency, hematological indicators: total bilirubin> 1.5 × ULN, ALT, AST> 2.5 × ULN; serum creatinine> 2 × ULN;
7. Those with a neutrophil count of less than 1.5 × 109 / L, or a platelet count of less than 100 × 109 / L, or an HGB of less than 90g / L;
8. Hepatitis B surface antigen, anti-HCV, anti-HIV or syphilis antibody positive;
9. Those who need to take valproic acid and drugs that can cause bone marrow depression during the application or research period;
10. pregnant or lactating women or those planning to become pregnant;
11. People with history of difficulty in drawing blood;
12. People with a history of bleeding disorders;
13. Subjects had a history of drug use or smoking and alcohol abuse within 6 months before enrollment;
14. Researchers do not consider it appropriate to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-10 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Tumor size | Four weeks after concurrent chemoradiotherapy, patients were then to receive three cycles of adjuvant temozolomide according to the standard 5-day schedule every 28 days. At the end of Cycle 3 (each cycle is 28 days)
  A tumor response was defned as a decrease of more than 30% of the largest tumor diameter or stable in Tumor volume

SECONDARY OUTCOMES:
Hormonal responses | Four weeks after concurrent chemoradiotherapy, patients were then to receive three cycles of adjuvant temozolomide according to the standard 5-day schedule every 28 days. At the end of Cycle 3 (each cycle is 28 days)
  Hormonal response as a 50% or more decrease in baseline hormone levels.

CONTACTS AND LOCATIONS:
Overall Officials: renzhi Wang, Dr., Study Director — pumch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burman P, Casar-Borota O, Perez-Rivas LG, Dekkers OM. Aggressive Pituitary Tumors and Pituitary Carcinomas: From Pathology to Treatment. J Clin Endocrinol Metab. 2023 Jun 16;108(7):1585-1601. doi: 10.1210/clinem/dgad098. PMID 36856733